CLINICAL TRIAL: NCT00996710
Title: Genomic Structural Variation in Cancer Susceptibility
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Cold Spring Harbor Laboratory (Other); Coriell Institute (Unknown); Weill Medical College of Cornell University (Other); University of Washington Center for Mendelian Genomics (Unknown)
Responsible Party: Sponsor
Other Study IDs: 09-068
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Colon Cancer; Germ Cell Cancer; Neuroblastoma; Rectal Cancer; Sarcoma
Keywords: Genome-wide; 09-068
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Neoplasms, Germ Cell and Embryonal; Neuroblastoma; Rectal Neoplasms; Sarcoma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood or saliva sample

SUMMARY:
This study will look for new types of gene changes that may be related to cancer in some patients. Some gene changes (mutations) are passed on from parents to offspring (child). Other gene changes are new and are seen for the first time in a child. They are not seen in the parent.

Some of these gene changes may cause cancers in the offspring. We will look for gene changes by studying patients with cancer their parents and family members without cancer. In this study, we will be able to find gene changes that occur in the cancer patient but not in the rest of the family. Knowing the role that new gene changes play in cancer risk may help us find people at a higher risk of getting cancer.

ELIGIBILITY:
Inclusion Criteria:

* Proband must have living unaffected biologic mother and father available and eligible for participation in the study with one of the following (both incident and prevalent cases will be collected):

  * Colorectal cancer diagnosed at or under the age of 50.
  * Breast cancer diagnosed at or under the age of 45.
  * Germ cell tumor diagnosed at or under the age of 40.
  * Pediatric cancer of any type diagnosed at or under the age of 21
  * Adult cancer or pre-neoplastic condition of any type diagnosed at or under the age of 40
  * Cancer at any age in 2 or more siblings suggestive of a genetic etiology, such as brothers with testicular germ cell tumor or sisters with breast cancer and ovarian cancer
* Parents:

  * Must be the biologic mother and biologic father of affected proband.
  * Must have (by self-report) no history of cancer other than non-melanomatous skin cancer or cervical cancer in situ except in the case of inclusion criteria #6..
  * In certain clinical situations, parent(s) with cancer may be included at the discretion of the Principal Investigator, if the Principal Investigator deems that the etiology of cancer in the parent(s) and proband are biologically unrelated.
* Sibling(s):

  * Must be age 18 or older and have same biologic parents as proband.

Exclusion Criteria:

* Known genetic mutation in proband or a family history that is indicative of hereditary cancer susceptibility.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The majority of eligible probands will be identified prospectively through the clinics of the Clinical Genetics, Medical Oncology and Pediatric Oncology Services of MSKCC by the patient's physician, the protocol investigator, or a research team member.
Sampling Method: Non-Probability Sample
Enrollment: 1275 (Actual)
Dates: Start 2009-10; Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To determine the frequency of de novo germline copy number variants (CNVs) in cancer affected probands using an ascertainment of "trios" consisting of cancer patients and their unaffected biologic parents | 2 years

SECONDARY OUTCOMES:
To explore the role of germline homozygosity in cancer susceptibility by determining the frequency and length of autozygous regions in patients with cancer | 2 years
  and mechanisms of Mendelian inheritance, such as autosomal recessive, autosomal dominant, and X-linked, which upon initial ascertainment may be difficult to decipher.

CONTACTS AND LOCATIONS:
Overall Officials: Zsofia Stadler, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org